CLINICAL TRIAL: NCT01504555
Title: Evaluation of the Diagnostic Utility of Serum Dexamethasone Measurements in the Overnight 1mg Dexamethasone Suppression Test in Patients Investigated for Cushing's Syndrome and Incidentalomas
Brief Title: Does Serum-DXM Increase Diagnostic Accuracy of the Overnight DXM Suppression Test in the Work-up of Cushing's Syndrome?
Acronym: DXM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/1810
Record Dates: First submitted 2011-11-15; First posted 2012-01-05 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Cushing's Syndrome; Adrenal Incidentalomas; Alcoholism; Obesity
Keywords: hypercortisolism, dexamethasone, alcoholism,obesity.
MeSH Terms: conditions — Cushing Syndrome; Adrenal incidentaloma; Alcoholism; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, saliva, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients under investigation for hypercortisolism: Patients undergoing routine evaluation for hypercortisolism at Haukeland University Hospital, Bergen, Norway, will be asked to participate.

SUMMARY:
Background: The evaluation for hypercortisolism includes an overnight 1mg dexamethasone (DXM) suppression test. An important shortcoming is the diagnostic specificity of only 80%, which is likely due to inter-individual differences in gut absorption or metabolism of DXM.

Study hypothesis: The investigators hypothesize that serum-DXM measurements will increase the diagnostic accuracy of the overnight DXM-test in the work-up of hypercortisolism.

Aims: The primary aim of this prospective study is to evaluate if serum-DXM measured simultaneously with serum-cortisol in morning samples could increase the diagnostic accuracy this diagnostic test. There are several secondary aims. One is to estimate the prevalence and causes of unusual DXM absorption or metabolism. The investigators will also evaluate the feasibility and diagnostic accuracy of salivary DXM. Moreover, the diagnostic accuracy of midnight salivary cortisol and cortisone, and urinary cortisol, will be evaluated and compared.

Design: Levels of DXM in morning serum following an overnight DXM-test will be analyzed in patients under evaluation for hypercortisolism (including incidentalomas). A cut-off level to identify inadequate DXM concentrations in serum to suppress endogenous cortisol production will be established based on the negative tests. This cut-off level will then be applied in a retrospective analysis of the diagnostic accuracy of DXM-tests. This prospective study has a blinded design as the DXM measurements are disclosed after the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Under investigation for hypercortisolism
* Able and willing to make informed consent

Exclusion Criteria:

* Use of systemic or local glucocorticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Haukeland University Hosptial, Bergen, Norway, under routine evaluation for hypercortisolism.Patients under evaluation for obeity at the overweight clinic, and Patients treated for alcohol abuse at the clinic for alcohol addicts at Haukeland University hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The difference (in percent) in false positive DXM-tests comparing the outcome of all tests with all tests excluding those with s-DXM below the the cut-off specified below. | 1 year
  The s-DXM cut-off will be defined a priori from ROC analysis on patients that inadequately suppress s-cortisol categorized as having Cushing's syndrome or being healthy.
  DXM, dexamethasone; DXM-test, short 1mg dexamethasone suppression test.

SECONDARY OUTCOMES:
Calculate the positive likelihood ratio [(1-sensitivity)/specificity] for the short DXM-test in the assessment of Cushing's syndrome (CS), after excluding those with s-DXM below the DXM cut-off specified in the primary endpoint. | 1 year
  Sensitivity = (Number of patients having CS with positive test / total number of patients with CS).
  Specificity = (Number of patients not having CS with negative test / total number of patients not having CS).
Calculate the negative likelihood ratio [(1-sensitivity)/specificity] for the short DXM-test in the assessment of Cushing's syndrome, after excluding those with s-DXM below the DXM cut-off specified in the primary endpoint. | 1 year
Calculate the positive likelihood ratio [(1-sensitivity)/specificity] for midnight salivary cortisol in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
Calculate the negative likelihood ratio [(1-sensitivity)/specificity] for midnight salivary cortisol in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
  A saliva cortisol cut-off level will be defined a priori from ROC analysis on all patients with and without Cushing's syndrome.
Calculate the positive likelihood ratio [(1-sensitivity)/specificity] for midnight salivary cortisone in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
  A saliva cortisone cut-off level will be defined a priori from ROC analysis on all patients with and without Cushing's syndrome.
Calculate the negative likelihood ratio [(1-sensitivity)/specificity] for midnight salivary cortisone in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
  A saliva cortisone cut-off level will be defined a priori from ROC analysis on all patients with and without Cushing's syndrome.
Identical to primary endpoint, but saliva-DXM measurements replace serum-DXM. | 1 year
Identical to primary endpoint, but saliva-DXM measurements replace serum-DXM, and saliva-cortisol replace serum-cortisol. | 1 year
Identical to primary endpoint, but saliva-DXM measurements replace serum-DXM and saliva-cortisone replace serum-cortisol. | 1 year
Calculate the positive likelihood ratio [(1-sensitivity)/specificity] for creatinine-adjusted cortisol in morning spot urine in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
  A cut-off level for creatinine-adjusted morning urine cortisol will be defined a priori from ROC analysis on all patients with and without Cushing's syndrome.
Calculate the negative likelihood ratio [(1-sensitivity)/specificity] for creatinine-adjusted cortisol in morning spot urine in the assessment of Cushing's syndrome. All study cases are included in this analysis. | 1 year
  A cut-off level for creatinine-adjusted morning urine cortisol will be defined a priori from ROC analysis on all patients with and without Cushing's Syndrome.
Compute a 95% confidence interval for morning s-DXM following overnight DXM-test in healthy subjects using parametric and non-parametric statistics. | 1 year
Quantitatively and qualitatively describe the characteristics of patients with false positive DXM-test and true negative DXM-test based on a standard questionnaire scoring patient history, symptoms and clinical features. | 1 year
  Parametric descriptive statistics
Evaluate the dexamethasone metabolism in patients with obesity | 1 year
  We are evaluating if overweight patients metabolise Dexamethasone in the same way as normal weighted patients, by looking at the s-dexamethasone and s-cortisol level the day after 1 mg overnight Dexamethason suppression test.
Evaluate the dexamethasone metabolism in patients with alcohol abuse | 1 year
  We are evaluating if patients with alcohol abuse metabolise dexamethasone in the same way as normal patients, by looking at the s-dexamethasone and s-cortisol level the day after 1 mg overnight dexamethason suppression test.

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Åstrøm Ueland, MD, Study Chair — Haukeland University Hospital
Locations (4):
- Norway (4):
  - Haukeland Universitetssykehus- Rusmedisinsk avdeling, Bergen
  - Haukeland Universitetssykehus- Endokrinologisk avdeling, Bergen
  - Institutt for farmakologi, Bergen
  - Haukeland University Hospital- Hormonlaboratory, Bergen

REFERENCES:
- [Background] Baid SK, Rubino D, Sinaii N, Ramsey S, Frank A, Nieman LK. Specificity of screening tests for Cushing's syndrome in an overweight and obese population. J Clin Endocrinol Metab. 2009 Oct;94(10):3857-64. doi: 10.1210/jc.2008-2766. Epub 2009 Jul 14. PMID 19602562
- [Background] Nieman LK, Biller BM, Findling JW, Newell-Price J, Savage MO, Stewart PM, Montori VM. The diagnosis of Cushing's syndrome: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2008 May;93(5):1526-40. doi: 10.1210/jc.2008-0125. Epub 2008 Mar 11. PMID 18334580
- [Background] Carroll TB, Findling JW. The diagnosis of Cushing's syndrome. Rev Endocr Metab Disord. 2010 Jun;11(2):147-53. doi: 10.1007/s11154-010-9143-3. PMID 20821267
- See also: Kortisol i spytt ved sykdom i binyrene — http://tidsskriftet.no/article/1502899
- See also: Spyttprøver til kortisolmåling — http://tidsskriftet.no/article/1501521
- See also: Endogent Cushing syndrom — http://tidsskriftet.no/article/1345319